CLINICAL TRIAL: NCT05028998
Title: The Impact of COVID-19-related Medication Assisted Treatment Policy Changes on Care and Outcomes for Patients With Opioid Use Disorder
Brief Title: COVID-19-Related Opioid Treatment Policy Evaluation
Acronym: COPE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Boston VA Research Institute, Inc. (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Boston University (Other); International Business Machines (IBM) (Industry)
Responsible Party: Sponsor
Other Study IDs: COVID-2020C2-11081
Record Dates: First submitted 2021-08-27; First posted 2021-08-31 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Opioid-use Disorder; Alcohol Use Disorder
Keywords: opioid use disorder, methadone, buprenorphine
MeSH Terms: conditions — Opioid-Related Disorders; Alcoholism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- Veterans with Opioid Use Disorder receiving care through the Veterans Health Administration: Pre-existing medical records data for these individuals will be part of our Aim 1 and Aim 2 large quantitative database.
  Additionally, we will be recruiting 30 of these individuals to participate in our Aim 3 qualitative interviews.
- Veterans with Alcohol Use Disorder receiving care through the Veterans Health Administration: Pre-existing medical records data for these individuals will be part of our Aim 1 and Aim 2 large quantitative database.
  We will not be recruiting any of these individuals for Aim 3 qualitative interviews.
- Patients with Opioid Use Disorder for whom Market Scan Medicaid Claims data is available: Pre-existing medical records data for these individuals will be part of our Aim 1 and Aim 2 large quantitative database.
  We will not be recruiting any of these individuals for Aim 3 qualitative interviews.
- Patients with Alcohol Use Disorder for whom Market Scan Medicaid Claims data is available: Pre-existing medical records data for these individuals will be part of our Aim 1 and Aim 2 large quantitative database.
  We will not be recruiting any of these individuals for Aim 3 qualitative interviews.
- Patients with Opioid Use Disorder for whom Market Scan Commercial Insurance Claims data is available: Pre-existing medical records data for these individuals will be part of our Aim 1 and Aim 2 large quantitative database.
  We will not be recruiting any of these individuals for Aim 3 qualitative interviews.
- Patients with Alcohol Use Disorder for whom Market Scan Commercial Claims data is available: Pre-existing medical records data for these individuals will be part of our Aim 1 and Aim 2 large quantitative database.
  We will not be recruiting any of these individuals for Aim 3 qualitative interviews.
- Patients with Opioid Use Disorder receiving care outside of Veterans Health Administration: We will be recruiting 30 of these individuals to participate in our Aim 3 qualitative interviews.
- Opioid Use Disorder Treatment Providers who provide treatment in the Veterans Health Administration: We will be recruiting 15 of these individuals to participate in our Aim 3 qualitative interviews.
- Opioid Use Disorder Providers who treat outside the Veterans Health Administration: We will be recruiting 15 of these individuals to participate in our Aim 3 qualitative interviews.
- Opioid Use Disorder Treatment and Policy Decision Makers: We will be recruiting 20 of these individuals to participate in our Aim 3 qualitative interviews.

SUMMARY:
Our nation is facing the COVID-19 pandemic during an ongoing opioid epidemic. Effective treatment for patients with opioid use problems involves a treatment method called Medication-Assisted Treatment, or MAT. In MAT, patients receive a medication that reduces cravings and withdrawal symptoms and can prevent overdose. Patients also receive counseling. Because the medications that are used in MAT are controlled substances, this treatment is subject to a number of federal regulations. The need for social-distancing during the pandemic would have made following these regulations very difficult for patients and their providers. Because of these difficulties, the federal government eased regulations in March 2020, making it easier for patients to receive MAT with fewer (if any) in-person visits for medication and counseling. Our team is studying the effects of these policy changes on the treatment that patients with opioid use disorder receive and on their outcomes. We are using both quantitative analyses of large, existing databases and qualitative analyses of interviews with patients, providers, and policy-makers to study these effects.

DETAILED DESCRIPTION:
The COVID-19 disease outbreak has occurred in the midst of a national opioid crisis, and poses significant risk for individuals with opioid use disorder (OUD). If existing in-person care delivery systems continued, patients would need to choose between risking exposure to the virus, or foregoing OUD treatment. Medication-assisted treatment (MAT), the gold-standard for treating OUD, involves daily medication (i.e., methadone or buprenorphine), close medication monitoring, and counseling sessions, all typically occurring in person. The medications used are schedule II and III controlled substances and are subject to greater federal regulations than medications for other substance use disorders (SUD), such as alcohol use disorder (AUD).3 To temper the impact of COVID-19 on OUD patients, in March 2020 the federal government temporarily, but dramatically, loosened MAT restrictions to expand treatment options, require fewer in-person visits, and prevent disruption to life-saving treatment.

This rapid shift in policy created a natural experiment, allowing for the evaluation of this MAT policy intervention on OUD patient care and outcomes. To examine the unknown effects of this intervention, we propose a mixed-methods, naturalistic experimental design involving quantitative analysis of large administrative and healthcare utilization datasets to evaluate the impact of MAT policy changes on patient care and outcomes. We will also compare OUD patient outcomes to those of AUD patients (analogue comparison group), for whom treatment was unaffected by MAT policy changes. We will then conduct interviews with patients, providers, and key MAT policy stakeholders, to understand perspectives on the impact of these COVID-19 related MAT policy changes on the lives and well-being of OUD patients, and guide policy decisions regarding whether or not to make these changes permanent. Given the general impact of the COVID-19 pandemic on patients and systems, we will compare outcomes for patients with OUD to analogue AUD patients, for whom there were no comparable medication policy changes in response to COVID-19.

Patients with OUD across three healthcare systems will be engaged in all steps of the research, including influencing the research design, assisting in determining key variables for Aims 1 and 2, collaborating in drafting our interview scripts for Aim 3, and assisting in interpreting our results and disseminating findings to patient stakeholders.

Aim 1. Using existing datasets, examine the effect of federal regulation changes on trends in delivery of MAT for OUD before and after pandemic onset, with a particular focus on prescription access, refills, and dosing schedules, as well as rates of in-person vs. telehealth medical and counseling visits.

Aim 2. Estimate the impact of the changes in OUD healthcare delivery on crucial patient outcomes (e.g., emergency department visits, detoxification, treatment retention, relapse, overdose, and mortality) by comparing patients with OUD vs. AUD (clinical analogue comparison group), across time (pre- and post-MAT policy changes).

Aim 3. Through in-depth, qualitative interviews and analyses, characterize patient, provider, and decision-maker perspectives on the impact of MAT policy changes in response to COVID-19 on patient access to MAT, health, functioning, and well-being.

Built-in reporting milestones will expedite data sharing to guide policy, provider, and patient decision-making as health care systems determine how to prepare for future pandemics, and post-COVID-19 pandemic care for OUD patients.

ELIGIBILITY:
Data for Aims 1 and 2 will be archival. Patients with OUD and their propensity score-matched AUD comparators will be included for Aims 1 and 2. No other patients from these larger datasets will be included.

In/exclusion below pertain to Aim 3 qualitative interviews:

Inclusion Criteria:

* VA patients with OUD who currently, or recently (within the past 6 months) receive(d) treatment for OUD from providers within Veterans Health Administration in the states of Massachusetts, Rhode Island, or New Hampshire.
* Non-Veteran patients with OUD (N=30) who currently, or recently (within the past 6 months) receive(d) treatment for OUD from providers outside Veterans Health Administration in the states of Massachusetts, Rhode Island, or New Hampshire.
* VA - OUD treatment providers who currently provide treatment for OUD within Veterans Health Administration, and have been a Veterans Health Administration provider of OUD treatment for at least one year in Massachusetts, Rhode Island, or New Hampshire.
* Non-VA OUD treatment providers who currently provide treatment for OUD outside of Veterans Health Administration, and have been a provider of OUD treatment for at least one year in Massachusetts, Rhode Island, or New Hampshire.
* OUD treatment and policy decision-makers who currently or recently (within past 6 months) hold/held positions within federal, state, or private organizations (e.g., Veterans Health Administration, SAMHSA) in which they are responsible for making and/or influencing significant decisions regarding the OUD treatment policy and/or the manner in which these are implemented.

Exclusion Criteria:

* Under 18
* Inability to speak fluent English
* Inability to provide a clear reporting of their experiences due to current influence of substances

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Veterans Health Administration and non-Veterans Health Administration (commercially and Medicaid-covered individuals) patients with OUD and their matched AUD comparators will be included in Aim 1 and 2 analyses. These represent archival claims (non-Veterans Health Administration data) and electronic health record data (Veterans Health Administration).
  The population for Aim 3 will include veterans who are current or recent patients of Veterans Health Administration, seeking/having received treatment for OUD at Veterans Health Administration; non-veterans seeking/having received treatment for OUD outside Veterans Health Administration; clinicians who treat patients with OUD within or outside Veterans Health Administration; and policy/decision-makers with expertise in opioid and OUD treatment policy.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Aim 1: Prescription medication access | January 2019-December 2019; April 2020-March 2021
  Medication prescription fills, In-person prescribing, Telehealth prescribing for OUD and AUD (clinical comparator)
Aim 1: Patient-provider encounter | January 2019-December 2019; April 2020-March 2021
  In-person counseling / psychotherapy, Telehealth counseling/ psychotherapy for OUD and AUD (clinical comparator)
Aim 2: Treatment retention/discontinuation | January 2019-December 2019; April 2020-March 2021
  Medication treatment retention, as measured by continuous and treatment, for patients with OUD and AUD (comparator)
Aim 2: Adverse outcomes | January 2019-December 2019; April 2020-March 2021
  Emergency Department visits, Detoxification treatment utilization, Overdose, Death, OUD/AUD Relapse for OUD and AUD (clinical comparator)
Aim 3: Semi-structured qualitative interview data from patients, providers, policy makers | January 2019-December 2019; April 2020-March 2021
  [Qualitative] Patient, provider, and policy-maker perspectives regarding OUD treatment and OUD treatment policies, practices, and implementation during COVID-19

CONTACTS AND LOCATIONS:
Locations (1):
- VA Boston Healthcare System, Boston, Massachusetts, United States